CLINICAL TRIAL: NCT04937998
Title: THE USE OF FRESH PRP VS HA IN THE TREATMENT OF OSTEOARTHRITIS OF THE PATELLOFEMORAL JOINT Randomized Controlled Clinical Trial
Brief Title: PRP Versus HA IN OSTEOARTHRITIS OF THE PATELLOFEMORAL JOINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-21
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: PRP; HA; Osteoarthritis; Autologous PRP; PRP injection; HA injection; injection treatment; Randomized controlled trial; Hyaluronic Acid; Platelet rich plasma
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded RCT in which one group of patients will be treated with 1 intra-articular injection of fresh PRP, and one group will be treated with 1 intra-articular injection of HA.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blinded randomized controlled trial with 1:1 allocation.Patient blinding will be provided during the injection treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous PRP injection (Experimental): This group of patients will be treated with single intra-articular injection of Autologous PRP.
  Interventions: Procedure: Autologous PRP injection
- HA injection (Active Comparator): This group of patients will be treated with single intra-articular injection of Hyaluronic Acid (HA)
  Interventions: Procedure: HA injection

INTERVENTIONS:
Procedure: Autologous PRP injection — Patients will be treated with a single injection of Autologous PRP (5 ml) in the knee joint affected by patellofemoral osteoarthritis
  Arms: Autologous PRP injection
Procedure: HA injection — Patients will be treated with a single injections of Hyaluronic Acid (5 ml) in the knee joint affected by patellofemoral osteoarthritis
  Arms: HA injection

SUMMARY:
The aim of the study is to compare the 12-month clinical outcomes of patients with patellofemoral osteoarthritis undergoing infiltrative treatment with fresh PRP and HA

DETAILED DESCRIPTION:
166 patients affected by patellofemoral osteoarthritis will be included in a double-blinded RCT. In this study one group of patients will be treated with 1 intra-articular injection of PRP (treatment arm) and one group will be treated with 1 intra-articular injection of HA (control arm). Patients will be followed-up with clinical evaluation at baseline and at 2.6.12 and 24 months. Questionnaires will be administered for clinical evaluations during the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 65;
2. Signs and symptoms of isolated patellofemoral osteoarthritis present in one or both knees;
3. Radiographic signs of isolated patellofemoral osteoarthritis (according to Iwano et al stage 1-3 classification) or chondropathy (assessed on MRI) with K-L grade of the other compartments ≤ 2. [PMID: 2302884 - PMID: 27979409] ;
4. Hemoglobin > 11 g/dl; Platelet count > 150,000 plt/mm3 (Recently performed CBC exam);
5. No clinically significant electrocardiographic alterations (Recently performed ECG).
6. Ability and consent of patients to actively participate in clinical follow-up;
7. Signature of informed consent.

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients who have undergone intra-articular infiltration of another substance within the previous 6 months;
3. Patients undergoing knee surgery within the previous 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with diabetes;
7. Patients with hematologic diseases (coagulopathies);
8. Patients on anticoagulant-antiaggregant therapy;
9. Patients with thyroid metabolic disorders;
10. Patients abusing alcoholic beverages, drugs or medications;
11. Body Mass Index > 35;
12. Patients who have taken NSAIDs in the 3 days prior to blood draw;
13. Patients with cardiovascular disease for which a 60 mL blood draw would be contraindicated;
14. Patients with a recently performed blood test with Hb< 11 g/dl and Platelets < 150,000 plt/mm3.
15. Previous treatment of patellar dislocation
16. Iwano score of grade 4.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
KOOS-Pain Score | 12 months
  KOOS-Pain Score is referred to a subscale of pain composed by 9 items. The score range considerate is 0-100.The score uses a 5-point Likert scale and each question is assigned a score from 0 to 4, where 0 indicates "no pain" and 4 "severe level of pain".

SECONDARY OUTCOMES:
IKDC-Subjective Score | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function.
KOOS-Pain Score | baseline, 2 month, 6 months , 24 months follow-up
  KOOS-Pain Score is referred to a subscale of pain composed by 9 items. The score range considerate is 0-100.The score uses a 5-point Likert scale and each question is assigned a score from 0 to 4, where 0 indicates "no pain" and 4 "severe level of pain".
Visual Analogue Scale (VAS) | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable".
EQ-VAS | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  EQ-VAS Is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
EQ-5D (EuroQoL) Current Health Assessment | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  EQ-5D is useful to evaluate the quality life of the patients
Tegner Activity Level Scale | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  Tegner activity level scale allows to know the level of physical activity carried out by the patients. All patients will indicate the type of sporting activity performed and its frequency.
Objective parameters- Range of Motion | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  Evaluation of the Range of Motion for comparative analysis.
Objective parameters - Circumferences | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis
Patient Acceptable Symptom State (PASS) | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
The Kujala Anterior Knee Pain Scale (AKPS) | baseline, 2 month, 6 months, 12 months , 24 months follow-up
  It's a 100-point scale consisting of 13 items with a score ranging from 5 to 10 points per item. A score of 0 points indicates the most severe limitation, while a score of 100 points indicates a normal situation.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694
- [Background] Cavallo C, Filardo G, Mariani E, Kon E, Marcacci M, Pereira Ruiz MT, Facchini A, Grigolo B. Comparison of platelet-rich plasma formulations for cartilage healing: an in vitro study. J Bone Joint Surg Am. 2014 Mar 5;96(5):423-9. doi: 10.2106/JBJS.M.00726. PMID 24599205
- [Background] deDeugd CM, Pareek A, Krych AJ, Cummings NM, Dahm DL. Outcomes of Patellofemoral Arthroplasty Based on Radiographic Severity. J Arthroplasty. 2017 Apr;32(4):1137-1142. doi: 10.1016/j.arth.2016.11.006. Epub 2016 Nov 15. PMID 27979409
- [Background] Assirelli E, Filardo G, Mariani E, Kon E, Roffi A, Vaccaro F, Marcacci M, Facchini A, Pulsatelli L. Effect of two different preparations of platelet-rich plasma on synoviocytes. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2690-703. doi: 10.1007/s00167-014-3113-3. Epub 2014 Jun 19. PMID 24942296